CLINICAL TRIAL: NCT03432000
Title: Study of the Links Between Perception of Temporal Order Judgment and Causality in Schizophrenic Spectrum Disorders
Brief Title: Links Between Perception of Temporal Order Judgment and Causality in Schizophrenia
Acronym: TOCAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator departure
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A03019-44
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This study consists in:
  * evaluate the links (correlation) between perception of temporal sequencing and perception of causality using an adapted experimental paradigm (Michotte paradigm) and to compare performance between healthy subjects and controls
  * investigate the existence of a correlation between these alterations and the peculiarities of the subjective experience of time (EAWE scale) in the group of subjects with schizophrenia
  The measures that will be realized are:
  * Performances of patients and controls on temporal task
  * Subjective alterations of time perception in patients with an adapted scale (EAWE)
  * Global symptomatology with PANSS (positive and negative symptom scale)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects with schizophrenia (Experimental): Performances on temporal task Subjective alterations of time perception in patients with an adapted scale (EAWE) Global symptomatology with PANSS (positive and negative symptom scale)
  Interventions: Other: Performances of patients and controls on temporal task
- healthy subjects (Sham Comparator): Evaluate the links (correlation) between perception of temporal sequencing and perception of causality using an adapted experimental paradigm (Michotte paradigm) and to compare performance between healthy subjects and controls Investigate the existence of a correlation between these alterations and the peculiarities of the subjective experience of time (EAWE scale) in the group of subjects with schizophrenia
  Interventions: Other: Performances of patients and controls on temporal task

INTERVENTIONS:
Other: Performances of patients and controls on temporal task — To carry out this work, we will rely on an experimental paradigm (derived from Michotte's paradigm) which makes it possible to explore the links between temporal sequencing and perception of causality, validated in the normal subject. subjective consequences of these alterations will be explored using a phenomenological-inspired clinical scale (EAWE time-scale items)

SUMMARY:
People with schizophrenia show disturbances in the perception of time. Among these alterations are the perturbations of the temporal order judgment. They are characterized by the fact that, as opposed to the general population, people with schizophrenia require a longer time interval between two successive stimuli to estimate which of the two events appeared first. If these alterations are now well documented, their consequences remain little explored. Among these consequences could however appear distortions of the judgment of causality (likely to underlie certain delusional interpretations) as well as a distressing experience of loss of the continuity of the lived experience (that could contribute to the alterations basic of self-awareness).

DETAILED DESCRIPTION:
The objective of our work lies in the study of the links between temporal sequencing, subjective perception of time and causality.

To carry out this work, the investigators will rely on an experimental paradigm (derived from Michotte's paradigm) which makes it possible to explore the links between temporal sequencing and perception of causality, validated in the normal subject. subjective consequences of these alterations will be explored using a phenomenological-inspired clinical scale (EAWE time-scale items)

ELIGIBILITY:
Inclusion Criteria:

Subjects with schizophrenia:

* Age from 18 to 45 years
* Diagnosis of schizophrenia according to DSM V criteria
* French mother tongue
* Psychotropic treatment unchanged during the month preceding the inclusion
* Stable symptomatology
* Normal or corrected visual acuity (> 0.8 at Snellen scale) and normal color vision
* Patients who gave informed consent to participate in the study

Control subjects (healthy volunteers):

* Age from 18 to 45 years
* Absence of neurological and psychiatric disorders
* French mother tongue

Exclusion Criteria:

* Recent addiction and abuse of cannabis or any other substance (according to DSM V criteria)
* Neurological disorders of vascular, infectious or neurodegenerative origin
* Taking somatic drugs with a cerebral or mental impact (eg corticosteroids)
* Disabling sensory disturbances, and in particular visual acuity
* Participation in a Neuro Cognitive Remediation Program
* Schizophrenia resistant to neuroleptic treatments
* Persons protected by law (pregnant women, minors, major under guardianship ...)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Comparison of the scores obtained by subjects with schizophrenia vs. the controls for the causal tasks, according to the delays between stimuli (stopping the moving launcher and appearance of the static object). | eight months
  Michotte paradigm: evaluate the links (correlation) between perception of temporal sequencing and perception of causality using an adapted experimental paradigm

SECONDARY OUTCOMES:
Comparisons of the scores obtained on the Time Experiment Rating Examination of Anomalous World Experience Scale (EAWE). | eight months
  Examination of Anomalous World Experience (EAWE ) scale:investigate the existence of a correlation between these alterations and the peculiarities of the subjective experience of time The E.A.W.E. consists of 6 dimensions (relation to space / relation to time / relation to others / language / atmospheric experience / existential orientation).The second domain only will be explored in our study Each item is both detailed, on a scale of 0 to 2 (0 for absent, 1 for present but with doubt, 2 for present, no doubt). The overall score of the sub-time scale thus ranges between 0 and 78.

CONTACTS AND LOCATIONS:
Overall Officials: MARTIN BRICE, Principal Investigator — CH LE VINATIER
Locations (1):
- Vial Veronique, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No